CLINICAL TRIAL: NCT02558920
Title: Important Food Sources of Fructose-Containing Sugars and Markers of Adiposity and Risk of Obesity: A Series of Systematic Reviews and Meta-Analyses of Controlled Trials and Prospective Cohort Studies
Brief Title: Meta-analyses of Food Sources of Fructose-Containing Sugars and Obesity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: John Sievenpiper (Other)
Collaborators: American Society for Nutrition (Other); The Physicians' Services Incorporated Foundation (Other); Canadian Diabetes Association (Other)
Responsible Party: Sponsor-Investigator, John Sievenpiper, Associate Professor, University of Toronto
Organization: University of Toronto (Other)
Other Study IDs: ASN-Sugars 2015
Record Dates: First submitted 2015-09-15; First posted 2015-09-24 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2018-12

CONDITIONS: Body Weight; Obesity; Overweight; Adiposity; Obesity, Abdominal
Keywords: Systematic review and meta-analysis; Evidence-based medicine (EBM); Evidence-based nutrition (EBN); Clinical practice guidelines; Clinical trials; Dietary sugars; Fructose; Sucrose; High fructose corn syrup; Isocaloric; Hypercaloric; Body weight; Prospective cohort studies
MeSH Terms: conditions — Body Weight; Obesity; Overweight; Obesity, Abdominal | interventions — Fructose; Sucrose; High Fructose Corn Syrup

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Fructose-containing Sugars — An intervention in which calories from food sources of fructose-containing sugars are substituted, added, subtracted, or replaced ad libitum in the diet
  Other Names: fructose, sucrose, high-fructose corn syrup (HFCS)

SUMMARY:
Sugars have been implicated in the epidemics of overweight and obesity. This view is supported by lower quality evidence from ecological observations, animal models, and select human trials. Higher level evidence from controlled trials and prospective cohort studies has been inconclusive. Whether sugars contribute to weight gain or increases in adiposity independent of their calories and whether important food sources of sugars other than SSBs are associated with a higher risk of overweight and obesity or weight gain remain unclear. To address the uncertainties, the investigators propose to conduct a series of systematic reviews and meta-analyses of the totality of the evidence from controlled trials and prospective cohort studies to distinguish the contribution of fructose-containing sugars and important food sources of sugars (SSBs, fruit, 100% fruit juice, cakes/sweets, yogurt, cereals, etc) from that of energy in the development of overweight and obesity. The findings generated by this proposed knowledge synthesis will help improve the health of consumers through informing evidence-based guidelines and improving health outcomes by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design

DETAILED DESCRIPTION:
Background: Sugars have emerged as one of the most important public health concerns. Attention has focused squarely on fructose-containing sugars (fructose, sucrose, high fructose corn syrup [HFCS], etc.). Collectively, these sugars have been indicted as drivers of the obesity epidemic and its and its downstream cardiometabolic complications. This special view rests on the unique metabolic and endocrine responses to fructose. Unlike glucose, fructose is thought to bypasses negative feedback control acting as an unregulated substrate for de novo lipogenesis and impair satiety signaling resulting in weight gain. In support of these mechanisms, animal models, low-quality ecological studies, and select human trials of overfeeding at levels of exposure far beyond population intakes have reported adverse metabolic effects of sugars. Higher level evidence from systematic reviews and meta-analyses of controlled trials, however, suggests that any effects of sugars are mediated by excess calories rather than the sugars per se. There is also evidence that not all food sources of these sugars are associated equally with obesity. While sugars-sweetened beverages (SSBs) have shown an adverse association with body weight, markers of adiposity and obesity, other important food sources of sugars such as fruit, 100% fruit juice, cereals, yogurts, and even cakes/sweets have shown either no association or a beneficial association. It remains unclear whether sugars contribute to weight gain or increases in adiposity independent of their calories and whether important food sources other than SSBs are associated with a higher risk of overweight and obesity.

Need for proposed research: High quality systematic reviews and meta-analyses of controlled trials and prospective cohort studies represent the highest level of evidence to support dietary guidelines and public health policy development. As dietary guidelines and public health policy have shifted toward food and dietary-pattern based recommendations, there is an urgent need for systematic reviews and meta-analyses comparing the role of different food sources of sugars in the development of overweight and obesity.

Objective: The investigators will conduct a series of American Society of Nutrition (ASN)-commissioned systematic reviews and meta-analyses to assess (1) the effect of different important food sources of sugars (e.g. SSBs, fruit, 100% fruit juice, yoghurt, cereals, cakes, pastries, sweets, etc.) at different levels of energy control on body weight and markers of adiposity in controlled trials and (2) their association with incident overweight/obesity and markers of adiposity in prospective cohort studies.

Design: Each systematic review and meta-analysis will be conducted according to the Cochrane Handbook for Systematic Reviews of Interventions and reported according to the Preferred Reporting Items for Systematic Reviews and Meta-Analyses (PRISMA).

Data sources: MEDLINE, EMBASE, and The Cochrane Central Register of Controlled Trials (Clinical Trials; CENTRAL) will be searched using appropriate search terms supplemented by hand searches of references of included studies.

Study selection: The investigators will include prospective cohort studies and controlled dietary trials. Prospective cohort studies will be included if they are >= 1-year duration and assess the relation of different sugars (total sugars, sucrose, fructose) or important food sources of added/free sugars (SSBs, pure fruit juice, cakes/sweets, cereals, yoghurt, etc.) with incident overweight/obesity or changes in markers of adiposity. Controlled (randomized and non-randomized) trials will be included if they are >= 2-weeks duration and assess the effect of fructose-containing sugars (fructose, sucrose, high fructose corn syrup, etc) from different food sources (e.g. SSBs, fruit, 100% fruit juice, yoghurt, cereals, cakes, pastries, sweets, etc.) on body weight or markers of adiposity. To allow for the separation of the effect of sugars from that of energy, 4 trial designs will be considered: (1) 'substitution' trials, in which fructose-containing sugars added to foods and beverages are compared with other macronutrient sources (usually starch or other sugars) under energy matched conditions; (2) 'addition' trials, in which fructose-containing sugars supplement a diet with excess energy compared to the same diet alone without the excess energy; (3) 'subtraction' trials, in which energy from fructose-containing sugars (usually in the form of sugars-sweetened beverages) is reduced by displacing it with water and/or no-calorie or low-calorie sweeteners or by eliminating it altogether from the background diet; and (4) 'ad libitum' trials, in which energy from fructose-containing sugars are freely replaced with other sources of energy without any strict control of either the study foods or the background diet.

Data extraction: Two or more investigators will independently extract relevant data and assess risk of bias using the Cochrane Risk of Bias Tool. All disagreements will be resolved by consensus. Standard computations and imputations will be used to derive missing variance data.

Outcomes: The primary outcome will be incidence of overweight/obesity in prospective cohort studies and body weight in controlled trials. Secondary outcomes will include measures of global adiposity (body weight [prospective cohort studies only], body mass index (BMI), and body fat) and measures of abdominal adiposity (waist circumference, waist-to-hip ratio, and visceral adipose tissue).

Data synthesis: Separate analyses will be conducted by level of energy control (substitution, addition, subtraction, ad libitum) and age (children, adults). Risk ratios will be pooled for incident overweight/obesity and mean differences for measures of global and abdominal adiposity using the generic inverse variance method. Random-effects models will be used even in the absence of statistically significant between-study heterogeneity, as they yield more conservative summary effect estimates in the presence of residual heterogeneity. Fixed-effects models will only be used where there is <5 included studies. Paired analyses will be applied for crossover trials. Heterogeneity will be assessed by the Cochran Q statistic and quantified by the I2 statistic. To explore sources of heterogeneity, the investigators will conduct sensitivity analyses, in which each study is systematically removed. If >=10 studies are available, then the investigators will also explore sources of heterogeneity by a priori subgroup analyses by sugar regulatory designation (added, naturally occurring), sugar food form (solid, liquid, or mixed), dose (=<10% energy, >10%), follow-up (=<10-years, >10-years), adjustment for adiposity, adjustment for energy, exposure assessment, dose, outcome ascertainment, risk of bias in prospective cohort studies and health status (metabolic syndrome/diabetes, overweight, normal weight), sugar type (sucrose, fructose, HFCS), sugar regulatory designation (added, naturally occurring), sugar food form (solid, liquid, or mixed), dose (=<10% energy, >10%), comparator (starch, fat, protein in substitution or ad libitum studies), baseline values, randomization, study design (parallel, crossover), energy balance (positive, neutral, negative), follow-up (=<8-weeks, >8-weeks), and risk of bias in controlled trials. Meta-regression analyses will assess the significance of categorical and continuous subgroups analyses. If >=10 studies are available, then publication bias will be investigated by inspection of funnel plots and formal testing using the Egger and Begg tests. If publication bias is suspected, then the investigators will attempt to adjust for funnel plot asymmetry by imputing the missing study data using the Duval and Tweedie trim and fill method.

Evidence Assessment: The certainty of the evidence for each outcome will be assessed using the Grading of Recommendations Assessment, Development and Evaluation (GRADE).

Knowledge translation plan: The results will be disseminated through interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Target audiences will include the public health and scientific communities with interest in nutrition, diabetes, obesity, and cardiovascular disease. Feedback will be incorporated and used to improve the public health message and key areas for future research will be defined. Applicant/Co-applicant Decision Makers will network among opinion leaders to increase awareness and participate directly as committee members in the development of future guidelines.

Significance: The proposed project will aid in knowledge translation related to the role of dietary fructose-containing sugars and important food sources of these sugars in the development of overweight and obesity, strengthening the evidence-base for guidelines and improving health outcomes by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

ELIGIBILITY:
Inclusion Criteria for controlled trials:

* Randomized and non-randomized controlled intervention studies in humans
* Oral fructose-containing sugars intervention
* Presence of a reduced fructose-containing sugars comparator in one of 4 energy controlled designs (substitution, addition, subtraction, or ad libitum)
* Diet duration >=2 weeks
* Viable outcome data

Inclusion Criteria for prospective cohort studies:

* Prospective cohort studies
* Duration >= 1 year
* Assessment of the exposure of food sources of fructose-containing sugars
* Ascertainment of viable outcome data by level of exposure

Exclusion Criteria for controlled trials:

* Observational studies or intervention studies with no control group
* IV or parenteral fructose-containing sugars intervention
* Lack of an adequate comparator (i.e. lack of a difference (<5 g) in fructose-containing sugars between the intervention and control diets)

Exclusion Criteria for prospective cohort studies:

* Ecological, cross-sectional, or retrospective observational studies
* Intervention studies

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All individuals, both children and adults, regardless of health status.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Incident overweight or obesity (prospective cohort studies) | Up to 20 years
  Incident overweight or obesity
Body weight (controlled trials) | Up to 20 years
  Body weight

SECONDARY OUTCOMES:
Global measures of adiposity with established clinical relevance - body weight (prospective cohort studies) | Up to 20 years
  Body weight
Global measures of adiposity with established clinical relevance - BMI (prospective cohort studies and controlled trials) | Up to 20 years
  Body mass index (BMI)
Global measures of adiposity with established clinical relevance - body fat (prospective cohort studies and controlled trials) | Up to 20 years
  Body fat
Abdominal measures of adiposity with established clinical relevance - waist circumference (prospective cohort studies and controlled trials) | Up to 20 years
  Waist circumference
Abdominal measures of adiposity with established clinical relevance - waist-to-hip ratio (prospective cohort studies and controlled trials) | Up to 20 years
  Waist-to-hip ratio
Abdominal measures of adiposity with established clinical relevance - Visceral Adipose tissue (prospective cohort studies and controlled trials) | Up to 2 years
  Visceral Adipose tissue (VAT)

CONTACTS AND LOCATIONS:
Overall Officials: John Sievenpiper, MD,PhD,FRCPC, Principal Investigator — University of Toronto
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Sievenpiper JL, de Souza RJ, Mirrahimi A, Yu ME, Carleton AJ, Beyene J, Chiavaroli L, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Kendall CW, Jenkins DJ. Effect of fructose on body weight in controlled feeding trials: a systematic review and meta-analysis. Ann Intern Med. 2012 Feb 21;156(4):291-304. doi: 10.7326/0003-4819-156-4-201202210-00007. PMID 22351714
- [Background] Sievenpiper JL, de Souza RJ, Cozma AI, Chiavaroli L, Ha V, Mirrahimi A. Fructose vs. glucose and metabolism: do the metabolic differences matter? Curr Opin Lipidol. 2014 Feb;25(1):8-19. doi: 10.1097/MOL.0000000000000042. PMID 24370846
- [Background] Sievenpiper JL, Chiavaroli L, de Souza RJ, Mirrahimi A, Cozma AI, Ha V, Wang DD, Yu ME, Carleton AJ, Beyene J, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Kendall CW, Jenkins DJ. 'Catalytic' doses of fructose may benefit glycaemic control without harming cardiometabolic risk factors: a small meta-analysis of randomised controlled feeding trials. Br J Nutr. 2012 Aug;108(3):418-23. doi: 10.1017/S000711451200013X. Epub 2012 Feb 21. PMID 22354959
- [Derived] Chiavaroli L, Cheung A, Ayoub-Charette S, Ahmed A, Lee D, Au-Yeung F, Qi X, Back S, McGlynn N, Ha V, Lai E, Khan TA, Blanco Mejia S, Zurbau A, Choo VL, de Souza RJ, Wolever TM, Leiter LA, Kendall CW, Jenkins DJ, Sievenpiper JL. Important food sources of fructose-containing sugars and adiposity: A systematic review and meta-analysis of controlled feeding trials. Am J Clin Nutr. 2023 Apr;117(4):741-765. doi: 10.1016/j.ajcnut.2023.01.023. Epub 2023 Feb 23. PMID 36842451